CLINICAL TRIAL: NCT00817804
Title: Cross-over Comparison of the V60 System to Other Bi-Level Noninvasive Ventilators for Pediatric Patients With Respiratory Failure or Respiratory Insufficiency
Brief Title: Cross-over Comparison of the V60 System to Other Bi-Level Noninvasive Ventilators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Respironics, California, Inc. (Industry)
Responsible Party: Dr. Steven Mink, Professor of Medicine, University of Manitoba, Winnipeg, Manitoba, Canada
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: V60-1050766VP v 2.3
Record Dates: First submitted 2009-01-03; First posted 2009-01-06 (Estimated); Results first posted 2009-08-12 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Respiratory Insufficiency; Respiratory Failure
Keywords: noninvasive ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- V60 then Conventional (Experimental): Study device first
  Interventions: Device: Use of the V60 Mask Ventilator
- Conventional then V60 (Experimental): Conventional device first
  Interventions: Device: Use of the V60 Mask Ventilator

INTERVENTIONS:
Device: Use of the V60 Mask Ventilator — The V60 Mask Ventilator used to provide noninvasive ventilation. It is compared to the patient's conventional ventilator in a cross-over study. The ventilator settings can range from CPAP to Pressure Support ventilation with values of IPAP and EPAP to match the conventional ventilation on which the patient had been placed.
  Other Names: V60 is the Philips V60 Ventilator

SUMMARY:
The purpose of this study is to compare a new noninvasive ventilator to existing ventilators already used for patient care.

DETAILED DESCRIPTION:
This study compares the Respironics California V60 Mask ventilator to conventional noninvasive ventilators in a cross-over study with the patient as his/her own control.

ELIGIBILITY:
Inclusion Criteria:

* Age > 7 years and < 18 years
* Weight > 20 kg (44 lbs)
* Respiratory failure or respiratory insufficiency
* Ability to cooperate with the investigators
* Designated adult able to provide Informed Consent

Exclusion Criteria:

* An endotracheal tube or tracheostomy in place
* Hemodynamically instability
* Prolonged apnea
* Inability to maintain the airway
* A recent history of cardiac and or respiratory arrest
* Acute hemorrhage
* Multiple organ system failure
* Undrained pneumothorax
* High risk for aspiration
* Metastatic or terminal cancer
* Do-not-resuscitate orders
* Inability to clear respiratory secretions
* Inability to fit a mask
* Facial surgery, trauma, or deformity
* Upper gastrointestinal or airway surgery
* Pregnancy
* Refractory delirium
* PaO2 < 50 mmHg on present settings
* Designee unable or unwilling to provide Informed Consent

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Mink, MD, Principal Investigator — University of Manitoba, Winnipeg, Manitoba, Canada
Locations (1):
- GF-221 Health Sciences Centre, Winnipeg, Manitoba, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitalized adult patients enrolled between Jan 17 and Mar 3, 2009.
Pre-assignment Details: Excluded if did not meet inclusion or did meet exclusion criteria.
Groups:
- V60 First: Experimental Study device (used as the experimental device) first in the cross-over study
- Conventional First: Experimental Study device (used as the experimental device) second in the cross-over study
Period: Overall Study
Arm/Group | V60 First | Conventional First
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V60 First | Conventional First | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 16.0 (0) | 11.5 (4.9) | 13.0 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Breathing Comfort
Description: Comfort on visual analog scale 0 - 100, 0 is best
Time Frame: 30 minutes
Population: Analysis was per protocol
Measure: Mean (Standard Error); unit: visual analog scale
Arm/Group | V60 First | Conventional First
Number analyzed (Participants) | 1 | 2
visual analog scale
  V60 | 10 (0) | 40 (14.1)
  Conventional | 33.3 (0) | 45 (7.1)

2. Secondary Outcome: Saturation of Arterial Oxygen
Time Frame: 30 minutes
Reporting Status: Not Posted, anticipated posting 2011-12
Measure: Number; unit: Percent

3. Secondary Outcome: Respiratory Rate
Description: Breathing rate in breaths per minute
Time Frame: 30 minutes
Reporting Status: Not Posted, anticipated posting 2011-12
Measure: Number; unit: Breaths per minute

4. Secondary Outcome: Minute Ventilation
Description: Liters per minute that the patient breathes
Time Frame: 30 minutes
Reporting Status: Not Posted
Measure: Number; unit: liters per minute

5. Secondary Outcome: Heart Rate
Description: Beats per minute that the patient's heart is beating
Time Frame: 30 minutes
Reporting Status: Not Posted
Measure: Number; unit: Beats per minute

6. Secondary Outcome: Blood Pressure
Description: Systolic and diastolic blood pressure
Time Frame: 30 minutes
Reporting Status: Not Posted
Measure: Number; unit: mm Hg

ADVERSE EVENTS:
Arm/Group | V60 First | Conventional First
Serious Adverse Events (participants affected / at risk) | 0 | 0
Other Adverse Events (participants affected / at risk) | 0 | 0

LIMITATIONS AND CAVEATS:
Terminated before 20 patients enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less